CLINICAL TRIAL: NCT00270062
Title: A Double-Blind, Placebo-Controlled Study to Determine Whether R-HuEPO Can Facilitate Presurgical Autologous Blood Donation in Patients With Low Hematocrit Levels
Brief Title: A Study to Evaluate the Safety of Epoetin Alfa and Its Effectiveness in Facilitating the Presurgical Collection of Blood From Anemic Patients for Possible Self-transfusion During and After Scheduled Joint Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005893
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-02

CONDITIONS: Anemia
Keywords: anemia; blood transfusion; epoetin alfa; erythropoietin; surgery; blood donation; blood
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety of epoetin alfa and its effectiveness in facilitating the presurgical collection of blood from anemic patients for possible self-transfusion during and after scheduled joint surgery and its effectiveness in reducing surgery-related transfusion requirements. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Major surgical procedures may require transfusion of several units of blood. Blood transfusions from other people may be associated with transfusion reactions that cause fever or infections such as hepatitis or AIDS that are carried (and donated) in blood. However, self-donations of blood may cause anemia in a patient who will be undergoing surgery a few weeks later. Previous research with epoetin alfa suggests that epoetin alfa increases the rate of red blood cell production and decreases anemia. This randomized, double-blind, placebo-controlled, multicenter study is designed to determine whether epoetin alfa in patients with low hematocrit (red blood cell percentage <39 percent) will stimulate the bone marrow to produce red blood cells and therefore increase a patient's ability to self-donate blood prior to major surgery for joint diseases. Patients will be randomly assigned to receive either 600 units of epoetin alfa per kilogram of body weight or matching placebo, injected into a vein on the first study day, and every 3 to 4 days thereafter for 21 days. Effectiveness will be determined by the number of units of self-donated blood collected, the number of units of donor blood used at the time of surgery, and the red blood cell percentages just before surgery. Safety evaluations including the incidence of adverse events, physical examinations, and clinical laboratory tests will be performed throughout the study. The study hypothesis is that patients treated with epoetin alfa will be able to donate more units of blood during the 3 weeks prior to surgery, will need fewer donor-donated units of blood, and will have a higher level of red blood cells than patients who receive placebo. 600 units of epoetin alfa per kilogram of body weight, or an equivalent volume of placebo, injected into a vein every 3 to 4 days for 21 days (6 doses) during the period before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery involving the joints, 25 to 35 days after starting epoetin alfa therapy
* having a hematocrit (percentage of red cells in the blood) of <=39%
* in good general health.

Exclusion Criteria:

* Patients with a history of any primary blood disease
* having a history of artery blockage in the heart, body or brain, a history of seizures, uncontrolled high blood pressure, or active inflammatory disease, (except osteoarthritis or rheumatoid arthritis)
* losing blood internally from the stomach or intestines or elsewhere in the body
* using of any cell toxic drug, drugs that suppress the immune system, or drugs known to influence red blood cell production (such as chemotherapy for cancer) within 1 month of therapy
* having a folate or vitamin B12 deficiency, iron-deficiency anemia, or a disease that destroys blood cells.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 1989-05; Study Completion 1991-07 (Actual)

PRIMARY OUTCOMES:
Number of units of blood self-donated; Number of donor-donated units of blood used; Total red blood cell volume; Total red blood cell production; Change in hemoglobin from baseline to after the final dose of study medication, but before surgery

SECONDARY OUTCOMES:
Total transfusion requirements at the time of surgery; incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to evaluate the safety of epoetin alfa and its effectiveness in facilitating the presurgical collection of blood from anemic patients for possible self-transfusion during and after scheduled joint surgery. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=677&filename=CR005893_CSR.pdf